CLINICAL TRIAL: NCT02916160
Title: Evaluation in Real Life Conditions of Sacubitril-valsartan Combination in Patients With Chronic Heart Failure and Sleep Apnea Syndrome
Brief Title: Sacubitril-valsartan and Heart Failure Patients : the ENTRESTO-SAS Study
Acronym: ENTRESTO696
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 9703
Record Dates: First submitted 2016-09-09; First posted 2016-09-27 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2020-07

CONDITIONS: Chronic Heart Failure; Sleep Apnea Syndrome
Keywords: Chronic Heart failure; Sleep Apnea Syndrome; Continuous Positive Airways Pressure; SACUBITRIL - VALSARTAN
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SACUBITRIL - VALSARTAN (Experimental): SACUBITRIL - VALSARTAN (formerly LCZ696, ENTRESTO®) is a new treatment of HF recently indicated class I, level B in the recent ESC guidelines 2016 on HF. It combines inhibitory prodrug neprilysin and valsartan.
  Interventions: Drug: SACUBITRIL - VALSARTAN (formerly LCZ696, ENTRESTO®)

INTERVENTIONS:
Drug: SACUBITRIL - VALSARTAN (formerly LCZ696, ENTRESTO®) — SACUBITRIL - VALSARTAN (formerly LCZ696, ENTRESTO®) is a new treatment of HF recently indicated class I, level B in the recent ESC guidelines 2016 on HF. It combines inhibitory prodrug neprilysin and valsartan.
  Other Names: LCZ696, ENTRESTO®

SUMMARY:
Chronic Heart Failure (CHF) is a frequent pathology burdened with mortality and significant morbidity. Sleep apnea syndrome (SAS) is frequently associated with CHF in 20% to 75% of cases. Treatment of SAS is however inconsistently associated with a decline in the morbidity and mortality. To date, the CHF medical treatments have been reported to be inconsistently efficient in the treatment of SAS.

SACUBITRIL-VALSARTAN (ENTRESTO®) is a new treatment of CHF recently indicated class I, level B in the recent European Society of Cardiology (ESC) guidelines 2016 on CHF. PARADIGM-HF trial demonstrated that morbidity and mortality can be improved with SACUBITRIL-VALSARTAN. In comparison to enalapril, it reduced the occurrence of cardiovascular death or hospitalisation for CHF by 20% with a 16% reduction in all-cause mortality.

The purpose of the research is the evaluation of SACUBITRIL-VALSARTAN combination in CHF patients presenting sleep apnea syndrome. A three months real life observational trial is performed. A measure of the Apnea Hypopnea Index is realised before and after 3 months of SACUBITRIL-VALSARTAN treatment. A concomitant evaluation of cardiological and quality of life parameters is realized.

DETAILED DESCRIPTION:
The Chronic Heart Failure (CHF) is a frequent pathology burdened with mortality and significant morbidity. Chronic HF provides almost 2% of health expenditure in developed countries, it is the largest expenditure item in the USA (34.8 billion dollars). In most developed countries, including France, mortality 1 year after diagnosis of chronic HF is 40%, it is 50% at 2 years, and over 70% at 4.5 years.

Sleep apnea syndrome (SAS) is frequently associated with HF in 20% to 75% of cases. The presence of an apnea syndrome is associated with a greater morbidity and mortality. Treatment of SAS is however inconsistently associated with a decline in the morbidity and mortality. To date, the CHF medical treatments have been reported to be inconsistently efficient in the treatment of SAS : 6 studies corresponding to a total of 67 patients and 5 types of molecules reported an incomplete effect on the central component of the Apnea Hypopnea Index (AHI) for these patients.

SACUBITRIL - VALSARTAN (ENTRESTO®) is a new treatment of HF recently indicated class I, level B in the recent ESC guidelines 2016 on HF. It combines inhibitory prodrug neprilysin and valsartan. After initial failures with neprilysin inhibition alone or dual neprilysin-angiotensin converting enzyme (ACE) inhibition, the PARADIGM-HF trial demonstrated that morbidity and mortality can be improved with the SACUBITRIL - VALSARTAN combination (formerly LCZ696). In comparison to the ACE inhibitor enalapril, sacubitril/valsartan reduced the occurrence of the primary end point (cardiovascular death or hospitalisation for HF) by 20% with a 16% reduction in all-cause mortality. These findings suggest that sacubitril/valsartan should replace an ACE inhibitor or angiotensin receptor blocker as the foundation of treatment of symptomatic patients (NYHA II-IV) with HF and a reduced ejection fraction.

The purpose of the research is the evaluation of SACUBITRIL-VALSARTAN in CHF patients presenting sleep apnea syndrome. We speculate that synchronously of a beneficial effect on heart failure, the SACUBITRIL-VALSARTAN combination could improve an associated SAS and in particular the central component of the AHI index.

After an exhaustive initial pre-therapeutic evaluation, the SACUBITRIL-VALSARTAN combination treatment is initiated for 3 months.

The pre-therapeutic evaluation includes cardiological and biological exams, quality of life questionaries and nocturnal ventilatory polygraphy.

Considering the results of the polygraphy, three groups of patients are identified:

* group 1 patients, characterized by a central AHI ≥5 / h and an obstructive AHI <15 / h,
* group 2 patients, characterized by an obstructive AHI ≥15 / h whatever is the central component. In this group of patient, a ventilator treatment with constant positive airway pressure or auto-servoventilation is started.
* group 3 patients, characterized by a central AHI < 5 / h and an obstructive AHI <15 / h.

After three months of treatment, the final evaluation includes cardiological and biological exams, quality of life questionaries for all the patient included in the trial. A nocturnal polygraphy is performed only in group 1 and 2 patients. For group 2 patients treated with a device, the observance to the device, the residual AHI device and the pressure device is measured.

ELIGIBILITY:
Inclusion Criteria:

* Age is greater than or equal to 18 years
* Patient with chronic heart failure (LVEF ≤ 45%).
* Written informed consent

Exclusion Criteria:

* Renal insufficiency (GF<30 milliliters/min)
* Pregnancy
* Allergy to one compound
* Personal history of angiooedema
* Hemodynamical instability
* Severe hepatopathy
* Current and not treated hyperkaliemia
* Prognosis < 6months
* Current CPAP or ASV treatment for Sleep Apnea Syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Changes in Apnea-Hypopnea Index as compared to baseline | 0 month to 3 months
  Changes in AHI as compared to baseline Measure of the apnea hypopnea index by a polygraphy performed before and after 3 months of treatment. The 2012 American Academy of Sleep Medicine recommendations are utilized in order to characterized apnea and hypopnea events, the central or obstructive or mixed phenotype

SECONDARY OUTCOMES:
Subject Global Assessment | 0 month to 3 months
NYHA Functional Class | 0 month to 3 months
Heart Rhythm | 0 month to 3 months
  physiological parameter
Systolic and diastolic Blood Pressure | 0 month to 3 months
  physiological parameter
Renal function as compared to baseline (Estimated GFR (eGFR) will be calculated using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula | 0 month to 3 months
  CKD-EPI formula
BNP (B-type Natriuretic Peptide) rates | 0 month to 3 months
  Biological parameter
Subject medications | 0 month to 3 months
Quality of life as measured by Minnesota Living with Heart Failure Questionary | 0 month to 3 months
  Questionaries
Quality of life as measured by EQ-5D-3L Questionary | 0 month to 3 months
  Questionaries
Epworth Sleepiness Scale | 0 month to 3 months
  Questionary
Pichot Fatigue Scale | 0 month to 3 months
  Questionary
Type of device used in group 2 patients | 0 month to 3 months
  CPAP or ASV device CPAP/ASV : continuous positive airway pressure / adaptive servo ventilation
CPAP/ASV compliance in group 2 patients | 0 month to 3 months
  CPAP/ASV compliance. Unit : number of hour per day using CPAP/ASV device
Historical of CPAP/ASV compliance in group 2 patients | 0 month to 3 months
  CPAP/ASV compliance. Unit : number of day with ≥3 hours in the past 6 months
Settings of CPAP/ASV device used in group 2 patients | 0 month to 3 months
  Settings of device
Type of mask used in group 2 patients | 0 month to 3 months
  Type of mask
Historical use of mask in group 2 patients | 0 month to 3 months
  Historical use of mask
Changes in AHI compared to Baseline in group 2 patients | 0 month to 3 months
  Changes in AHI compared to Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BOURDIN, MD,PhD, Study Director — University Hospital, Montpellier
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux, Pessac
  - Pôle médical spécialisé MSP, Béziers
  - CHU Béziers, Béziers
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jaffuel D, Molinari N, Berdague P, Pathak A, Galinier M, Dupuis M, Ricci JE, Mallet JP, Bourdin A, Roubille F. Impact of sacubitril-valsartan combination in patients with chronic heart failure and sleep apnoea syndrome: the ENTRESTO-SAS study design. ESC Heart Fail. 2018 Jun;5(3):222-230. doi: 10.1002/ehf2.12270. Epub 2018 Feb 22. PMID 29469206
- [Result] Jaffuel D, Nogue E, Berdague P, Galinier M, Fournier P, Dupuis M, Georger F, Cadars MP, Ricci JE, Plouvier N, Picard F, Puel V, Mallet JP, Suehs CM, Molinari N, Bourdin A, Roubille F. Sacubitril-valsartan initiation in chronic heart failure patients impacts sleep apnea: the ENTRESTO-SAS study. ESC Heart Fail. 2021 Aug;8(4):2513-2526. doi: 10.1002/ehf2.13455. Epub 2021 Jun 8. PMID 34102018